CLINICAL TRIAL: NCT06305871
Title: Clinical Study of Ultrasound-guided Radiofrequency Ablation in the Treatment of Refractory Hyperthyroidism
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhang Bo (Other)
Responsible Party: Sponsor-Investigator, Zhang Bo, Chief Physician, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-NHLHCRF-YYPPLC-ZR-09
Record Dates: First submitted 2024-02-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Hyperthyroidism/Thyrotoxicosis
Keywords: Hyperthyroidism; Ultrasound-guided ablation
MeSH Terms: conditions — Hyperthyroidism; Thyrotoxicosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ablation group (Experimental): Patients with hyperthyroidism undergoing ultrasound-guided ablation
  Interventions: Procedure: Ablation therapy

INTERVENTIONS:
Procedure: Ablation therapy — Ablative treatment of hyperthyroidism

SUMMARY:
Hyperthyroidism is an endocrine disease with a high incidence rate, and some patients are difficult to effectively control the condition after long-term drug treatment, and the disease recurs, forming refractory hyperthyroidism. The search for a new safe, effective and minimally invasive treatment has become a research hotspot. Ultrasound-guided radiofrequency ablation is a hot spot in clinical research due to its advantages of low trauma, high safety, precise inactivation of lesions, and multiple ablation. However, there is no unified standard for the number and scope of ablation in the treatment of refractory hyperthyroidism by radiofrequency ablation, and there is a lack of data on the effectiveness and safety of the treatment with large samples and long-term effects. Therefore, how to establish a standardized treatment strategy and appropriate plan for ablation of refractory hyperthyroidism based on clinical practice is an urgent problem to be solved. The purpose of this study was to prospectively include refractory hyperthyroidism for ultrasound-guided radiofrequency ablation, and to evaluate the efficacy and safety of hyperthyroidism ablation by comparing the changes in symptoms and signs, serology, and imaging of patients before and after ablation. The relevant factors affecting the efficacy of ablation were analyzed and the most appropriate ablation scope was determined. Radiofrequency ablation was retrospectively compared with traditional surgery and 131I treatment, and the near- and medium-term treatment effects, incidence of adverse reactions and complications, as well as the economic benefits and sociopsychological differences of the three treatment methods were compared.

The expected outcome of this study is to establish a research cohort of hyperthyroidism ablation based on a large sample population, and to establish the most appropriate and effective regimen for radiofrequency ablation of refractory hyperthyroidism compared with traditional surgery and 131I treatment with safety and near- and medium-term efficacy. The Department of Ultrasound Medicine of China-Japan Friendship Hospital has accumulated rich experience in the ablation treatment of benign and malignant thyroid nodules and hyperthyroidism, and has completed more than 200 cases of thyroid ablation in the past two years. Under the leadership of Professor Zhang Bo, the research team of this project has conducted a number of clinical studies on the ultrasound diagnosis and treatment of thyroid diseases, presided over and participated in more than 20 national, provincial and university-level scientific research courses, and the first author or corresponding author wrote more than 70 articles in related fields, which laid a solid research foundation for the conduct of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Poor effect and recurrence after medical standard treatment
2. serious adverse reaction to drug treatment
3. poor effect of iodine-131 treatment
4. Patients who wish to undergo ablation surgery to shorten the duration of treatment and improve symptoms
5. Moderate to severe active Graves ophthalmopathy
6. Second trimester patients

Exclusion Criteria:

1. Poor general condition
2. early and late pregnancy
3. The retrosternal thyroid or thyroid gland is mostly behind the sternum
4. Incomplete function of one vocal cord
5. severe coagulation dysfunction
6. Malignant exophthalmia
7. Adolescent patients
8. Patients requiring urgent relief of symptoms of oppression.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Discontinuation rate | two years
  Discontinuation rate in patients with hyperthyroidism ablation for six months after surgery
Recurrence rate | two years
  Recurrence rate in patients with hyperthyroidism ablation half a year after discontinuation of the drug

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan friendship hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No